CLINICAL TRIAL: NCT01055340
Title: A Randomized Clinical Trial to Study Ketogenesis and Glucose-Dependent Insulin Secretion Methodologies in Healthy Male Subjects
Brief Title: A Study That Will Evaluate Ketogenesis and Glucose-Dependent Insulin Secretion Methodologies in Healthy Male Subjects (MK-0000-159)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-159; 159; 2010_506
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
Keywords: Ketogenesis; Glucose-Dependent Insulin Secretion; Graded Glucose Infusion; Oxyntomodulin
MeSH Terms: conditions — Obesity | interventions — Oxyntomodulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment sequence 1 (Experimental): OXM 3.0 pmol/kg/min - OXM 0.6 pmol/kg/min - Placebo
  Interventions: Drug: Oxyntomodulin (OXM); Drug: Comparator: Oxyntomodulin (OXM); Drug: Comparator: Placebo [ hemaccel-containing saline]
- Treatment sequence 2 (Experimental): OXM 0.6 pmol/kg/min - Placebo - OXM 3.0 pmol/kg/min
  Interventions: Drug: Oxyntomodulin (OXM); Drug: Comparator: Oxyntomodulin (OXM); Drug: Comparator: Placebo [ hemaccel-containing saline]
- Treatment sequence 3 (Experimental): Placebo - OXM 3.0 pmol/kg/min - OXM 0.6 pmol/kg/min
  Interventions: Drug: Oxyntomodulin (OXM); Drug: Comparator: Oxyntomodulin (OXM); Drug: Comparator: Placebo [ hemaccel-containing saline]
- Treatment sequence 4 (Experimental): OXM 3.0 pmol/kg/min - Placebo - OXM 0.6 pmol/kg/min
  Interventions: Drug: Oxyntomodulin (OXM); Drug: Comparator: Oxyntomodulin (OXM); Drug: Comparator: Placebo [ hemaccel-containing saline]
- Treatment sequence 5 (Experimental): Placebo - OXM 0.6 pmol/kg/min - OXM 3.0 pmol/kg/min
  Interventions: Drug: Oxyntomodulin (OXM); Drug: Comparator: Oxyntomodulin (OXM); Drug: Comparator: Placebo [ hemaccel-containing saline]
- Treatment sequence 6 (Experimental): OXM 0.6 pmol/kg/min - OXM 3.0 pmol/kg/min - Placebo
  Interventions: Drug: Oxyntomodulin (OXM); Drug: Comparator: Oxyntomodulin (OXM); Drug: Comparator: Placebo [ hemaccel-containing saline]

INTERVENTIONS:
Drug: Oxyntomodulin (OXM) — Single infusion of OXM 3.0 pmol/kg/min by IV
Drug: Comparator: Oxyntomodulin (OXM) — Single infusion of OXM 0.6 pmol/kg/min by IV
Drug: Comparator: Placebo [ hemaccel-containing saline] — Single Placebo infusion of hemaccel-containing saline by IV

SUMMARY:
This study will test the hypotheses that a single dose of oxyntomodulin (OXM) will be neutral or better than placebo in lowering ambient glucose levels during a graded glucose infusion (GGI) and that a single dose of OXM will lead to a statistically significant increase in the sum of the plasma βOHB + AcAc levels compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject is judged to be in good health based on medical history, physical examination, and laboratory safety tests
* Subject has a Body Mass Index of ≥27 kg/m^2 and ≤35 kg/m^2 and weighs ≥70 kg at the prestudy (screening) visit
* Subject has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months
* Subject is willing to avoid strenuous physical activity (weight lifting, running, bicycling, etc.) for the duration of the study

Exclusion Criteria:

* Subject is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit
* Subject has a history of stroke, chronic seizures, or major neurological disorder
* Subject has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* Subject has irritable bowel disease, or recurrent occurrences of nausea, vomiting, diarrhea, or abdominal pain
* Subject has a history of hypertension requiring treatment
* Subject has a history of cancer
* Subject has history of diabetes, or family history of diabetes mellitus
* Subject has a history of hypersensitivity to OXM or hemaccel

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Ambient plasma glucose concentration during the GGI | Last 160 minutes of OXM/placebo infusion
plasma βOHB + AcAc concentrations | First 300 minutes of OXM/placebo infusion

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Shankar SS, Shankar RR, Mixson LA, Miller DL, Pramanik B, O'Dowd AK, Williams DM, Frederick CB, Beals CR, Stoch SA, Steinberg HO, Kelley DE. Native Oxyntomodulin Has Significant Glucoregulatory Effects Independent of Weight Loss in Obese Humans With and Without Type 2 Diabetes. Diabetes. 2018 Jun;67(6):1105-1112. doi: 10.2337/db17-1331. Epub 2018 Mar 15. PMID 29545266
- [Derived] Shankar SS, Shankar RR, Mixson LA, Miller DL, Chung C, Cilissen C, Beals CR, Stoch SA, Steinberg HO, Kelley DE. Linearity of beta-cell response across the metabolic spectrum and to pharmacology: insights from a graded glucose infusion-based investigation series. Am J Physiol Endocrinol Metab. 2016 Jun 1;310(11):E865-73. doi: 10.1152/ajpendo.00527.2015. Epub 2016 Apr 12. PMID 27072496